CLINICAL TRIAL: NCT06053437
Title: Prognostic Indicators in Pituitary Adenoma Surgery: a Comprehensive Analysis of Surgical Outcomes and Complications.
Acronym: Hyp'Op
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, DEMARQUET Lea, Principal Investigator, Central Hospital, Nancy, France
Other Study IDs: 2022PI198
Record Dates: First submitted 2023-02-03; First posted 2023-09-25 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Pituitary Adenoma; Surgery-Complications
Keywords: transsphenoidal surgery; pituitary adenoma; post-operative complications
MeSH Terms: conditions — Pituitary Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hyp'Op Cohort: The 'HYP'OP' cohort comprises patients who underwent endoscopic endonasal surgery (EES) for pituitary adenoma during a 10-year period spanning from January 2012 to June 2022 at the Nancy University Hospital. Post-operative hospitalization in our endocrinology department is part of the standard care protocol, which also includes a systematic reevaluation 4 -6 months following the surgical intervention.

SUMMARY:
Predicting the outcome of pituitary surgery, particularly the risk of complications, is a critical determinant in selecting the appropriate treatment modality for patients. To date, only a limited number of risk factors have been identified for complications following pituitary surgery, including tumor size, younger age, and previous surgical intervention. Furthermore, existing studies have demonstrated that prolactin levels can serve as a surrogate marker for assessing pituitary function, specifically revealing associations between elevated prolactin levels and anterior pituitary insufficiencies.

In a retrospective study on the "HYP'OP" cohort, the aim of the study is to identify predictive factors for both surgical outcomes and complications.

ELIGIBILITY:
Inclusion Criteria:

* Transsphenoidal pituitary surgery at Nancy University Hospital (France) between 2012 and 2022 for a pituitary adenoma.

Exclusion Criteria:

* No 4 month evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients having undergone transsphenoidal pituitary surgery at Nancy University Hospital (France) between 2012 and 2022 for a pituitary adenoma are to be included.
Sampling Method: Non-Probability Sample
Enrollment: 211 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Risk factors associated with complications | Within 6 months after surgery
  Risk factors associated with complications arising from surgery, specifically targeting the incidence of de-novo, clinically significant pituitary insufficiencies

SECONDARY OUTCOMES:
Factors predictive of the 'success' of surgery | Within 6 months after surgery
  Patients were stratified into groups based on surgical indications. The first group consisted of non-secreting, non-compressive adenomas without preoperative insufficiency or hyperprolactinemia, with success defined as absence of new insufficiency and no MRI-detected residual tissue. The second group was similar to the first but included disconnection hyperprolactinemia, and success was defined by the absence of new insufficiency and hyperprolactinemia regression. The third group involved non-secreting adenomas with at least one preoperative axis deficiency, irrespective of hyperprolactinemia, with success defined as restoration of at least one deficient axis without new insufficiency. The fourth group included secreting adenomas, with success defined as hypersecretion regression. The fifth group involved adenomas operated on for their compressive effect on the optic pathways, with or without hyperprolactinemia, and success was defined as no compression observed on follow-up MRI.
Is immediate postoperative hypoprolactinemia predictive of the onset of a new, clinically significant hormonal insufficiency? | Within 6 months after surgery
  patients were stratified into four groups based on immediate postoperative prolactin levels: Group 1 consisted of severe hypoprolactinemia; Group 2 included moderate hypoprolactinemia; Group 3 involved normal prolactin levels, defined by prolactin levels between 5 and 20 ng/ml; and Group 4 comprised hyperprolactinemia, defined by prolactin levels > 20 ng/ml. It should be noted that these instances of hyperprolactinemia are theoretically all disconnection hyperprolactinemias, as patients with lactotroph adenomas were excluded from this analysis. Patients under treatment for hyperprolactinemia were also excluded.

OTHER OUTCOMES:
Is hypoprolactinemia at the 4-month follow-up is correlated with the number of affected pituitary axes? | Within 6 months after surgery
  Patients were stratified into four groups using the same criteria as outlined in Outcome 3.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Régional Universitaire de Nancy, Nancy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Riley G, Scheyer N, Klein M, Merlot I, Guerci B, Jeanbert E, Demarquet L. Prognostic indicators in pituitary adenoma surgery: a comprehensive analysis of surgical outcomes and complications. Front Endocrinol (Lausanne). 2024 Jan 11;14:1327404. doi: 10.3389/fendo.2023.1327404. eCollection 2023. PMID 38274233